CLINICAL TRIAL: NCT00000259
Title: Sevoflurane vs Nitrous Oxide Inhalation at Subanesthetic Concentrations
Brief Title: Sevoflurane vs Nitrous Oxide Inhalation at Subanesthetic Concentrations - 11
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double
Other Study IDs: NIDA-08391-11; R01DA008391 (NIH); R01-08391-11
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: sevoflurane; nitrous oxide; subjective effects; healthy volunteer
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Nitrous Oxide; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Placebo (Placebo Comparator): Subject inhales no drug (100% oxygen)
  Interventions: Other: Placebo
- 0.3% sevoflurane (Active Comparator)
  Interventions: Drug: 0.3 % Sevoflurane
- 0.6% sevoflurane (Active Comparator)
  Interventions: Drug: 0.6% Sevoflurane
- 15% Nitrous oxide (Active Comparator)
  Interventions: Drug: 15 % Nitrous oxide
- 30% Nitrous oxide (Active Comparator)
  Interventions: Drug: 30% Nitrous oxide

INTERVENTIONS:
Drug: 15 % Nitrous oxide
  Arms: 15% Nitrous oxide
Drug: 0.3 % Sevoflurane
  Arms: 0.3% sevoflurane
Drug: 30% Nitrous oxide
  Arms: 30% Nitrous oxide
Drug: 0.6% Sevoflurane
  Arms: 0.6% sevoflurane
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to conduct experiments to examine subjective and reinforcing effects of nitrous oxide. Mood altering and psychomotor effects will be tested on non-drug abusers and preference procedures will be used to assess reinforcing effects. Comparisons between nitrous oxide, opiates, and benzodiazepine antagonists will be made. To examine sevoflurane versus isoflurane inhalation at subanesthetic concentrations on mood, pain, and psychomotor performance.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 1996-08; Primary Completion 1997-11 (Actual); Study Completion 1997-11 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 30 min of inhalation
  Subjects underwent a 3 min cold immersion test at 30 min of inhalation and then provided response to pain intensity questionnaire
Psychomotor performance | Baseline, 5 min of inhalation; 5, 30, 60 minutes recovery
  Subjects underwent psychomotor testing at baseline, during inhalation, and during recovery post inhalation
Cognitive performance | Baseline, every 5 min during inhalation, 5, 30, & 60 min during recovery
  Subject underwent memory, sedation, visual analog, and drug effects testing

CONTACTS AND LOCATIONS:
Overall Officials: James Zacny, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Anesthesia & Critical Care, Chicago, Illinois, United States

REFERENCES:
- [Background] Anesthesiology. 1997 (in press).